CLINICAL TRIAL: NCT01199497
Title: Multicenter Clinical Trial Phase III, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Fixed Dose Combination of Diphenhydramine + Pseudoephedrine + Dropropizine in the Control of Cough and the Relief of Nasal Symptoms in Subjects Above 12 Years of Age, Suffering From Non-productive Cough and Acute Rhinitis.
Brief Title: Study to Evaluate the Efficacy and Safety of Fixed Dose Combination of Diphenhydramine + Pseudoephedrine + Dropropizine in the Control of Cough and the Relief of Nasal Symptoms, Suffering From Non-productive Cough and Acute Rhinitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-NTS-03(08/10)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Nasal Congestion; Cough
Keywords: cough, acute rhinitis, nasal congestion, common cold, nasal symptoms, children.; Nasal congestion and non-productive cough, with or without associate other nasal and extranasal symptoms.
MeSH Terms: conditions — Nasal Obstruction; Cough; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Fixed dose combination of diphenhydramine + dropropizine + pseudoephedrine (Notuss® syrup).
  Interventions: Drug: Group 1
- Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Group 2

INTERVENTIONS:
Drug: Group 1 — fixed dose combination of diphenhydramine + dropropizine + pseudoephedrine (Notuss® syrup).
  Arms: Group 1
Drug: Group 2 — placebo
  Arms: Group 2

SUMMARY:
Multicenter clinical trial, phase III, controlled by active medicine, double-blind, randomized, enroll 208 subjects, above 12 years old, that suffer acute inflammation upper airway characterized by non-productive cough, daytime/nighttime, with duration for at least 3 and no more than 5 consecutive days (without systemic/topic use of medication during this period) followed by nasal congestion, with or without associate other nasal symptoms (sneezing, runny nose, nasal itching and/or mouth breathing). The subjects will be allocated in 2 parallel groups, and will receive the medicines of study, according of the randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 12 years old, of both sexes;
2. Clinical condition compatible with acute rhinitis accompanied by nasal congestion;
3. Non-productive cough, daytime and/or nighttime with at least 3 and up 5 consecutive days in duration;
4. Score greater than or equal to 3 points on the cough severity score (As per item 4.1.2);
5. Score greater than or equal to 2 points on the nasal congestion severity score (As per item 4.1.3);
6. If necessary, ICF signed by a parent/representant, or in case the patient over 18 years old, his own signature;
7. Patient and/or representant capacity, according to investigator evaluation, for compliance at the treatment and protocol requirements, fulfilling the regular visits;

Exclusion Criteria:

1. Non-productive cough with purulent smear, fever (axilar temperature superior than 37,8°C/100°F), purulent runny nose and other signs and symptoms of bacteria infection of upper and lower airways at 7 days before the screening/randomization visit;
2. Septal deviation level III (in any region and any nasal cavity) and/or nasal polyps or other determinants conditions of nasal congestion;
3. Previous diagnosis of asthma;
4. Female patients with positive b-HCG;
5. Patients under treatment for chronic allergy;
6. Presence of purulent or mucupurulent secretion, nasal vault or mal formations (cleft lip or cleft nasolabial corrected or not) in nasal vestibule;
7. Current use of systemic antibiotics for any reason;
8. Use of prohibited medicine within the prescribed period before V0 as shown in item 9.3 of this protocol;
9. Participation in last one year of clinical protocols;
10. Any psychiatric diseases, including major depression;
11. Presence of mental retardation from any cause;
12. Diagnosis of renal or hepatic failure;
13. History of hypersensitivity to any component of the study drugs;
14. Relatives of sponsor´s or study site´s employee;
15. Current evidence of clinically significant diseases: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrine, psychiatric, autoimmune, pulmonary, or another disease that block the patient participation;
16. Patient or parent/representant with a history of lack of compliance to treatment or previous treatment protocols;
17. Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the patient or interfere with the endpoints of study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy criteria | baseline and week 24
  The changes of lung function parameter: pre-bronchodilator forced expiratory volume in first second (FEV1) including baseline and 24th week.

SECONDARY OUTCOMES:
Secondary efficacy criteria | baseline, week 8, 16 and 24
  Changes in forced expiratory volume in first second (FEV1).